CLINICAL TRIAL: NCT07264335
Title: A Randomized, Open-Label, Parallel-Group Clinical Study to Evaluate the Bioavailability and Safety of Subcutaneous SHR-1819 Injection Administered Using Different Injection Devices in Healthy Subjects
Brief Title: A Study on the Bioavailability of SHR-1819 Injection Administered Subcutaneously Using Different Injection Devices in Healthy Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Hengrui Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1819-105
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prefilled Syringe (PFS) Group (Experimental)
  Interventions: Drug: SHR-1819 Injection
- Artificial Intelligence (AI) Group (Experimental)
  Interventions: Drug: SHR-1819 Injection

INTERVENTIONS:
Drug: SHR-1819 Injection — SHR-1819 injection.

SUMMARY:
This study is a randomized, parallel-group, open-label Phase I clinical trial designed to compare the bioavailability and safety of subcutaneous SHR-1819 injection administered via different injection devices in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Understanding the research procedures and methods, being able to complete the research in accordance with the procedure requirements, and sign the informed consent;
2. The age on the date of signing the informed consent must be ≥18 years old and ≤55 years old;
3. Body mass index (BMI) at screening period must be ≥19.0 kg/m2 and <26.0 kg/m2, weight of male must≥ 50.0 kg and <80.0 kg;
4. The subjects and their female partners are willing to have no reproductive plan from signing the informed consent to 3 months after the last administration of the study drug, and voluntarily take effective contraceptive measures and do not plan to donate sperm or ovum.

Exclusion Criteria:

1. History of the following diseases or treatments: (1) Receipt of a live-attenuated vaccine within 1 month prior to screening or planned receipt during the study; (2) Previous participation in a clinical trial involving any investigational product (drug or device) within 3 months before screening; (3) History of food or drug allergy or atopic allergic disease (asthma, urticaria);
2. Any one of the following tests at Screening period or Baseline period: (1) Human immunodeficiency virus antibody (HIV-Ab), syphilis serological examination, hepatitis B virus surface antigen (HBsAg), hepatitis C virus antibody (HCV-Ab) positive; (2) Exclude individuals who have experienced severe trauma or undergone major surgery within the past 6 months, or who plan to undergo surgery during the trial period;
3. General situation: (1) Have a history of drug use or drug abuse; (2) Investigators, site staff, or any other individuals directly involved in the conduct of the protocol;
4. Subjects who are considered by the investigator to have any other factors which are not suitable for participating in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Area under the serum concentration versus time curve from time zero to the real time of last measurable concentration (AUClast). | Day 1 - Day 71.
Peak concentration (Cmax) | Day 1 - Day 71.
  Pharmacokinetic parameters of multiple-site subcutaneous injection of SHR-1819.

SECONDARY OUTCOMES:
SHR-1819 Anti-Drug Antibodies (ADA) | Day1; Day22 ; Day43; Day71.
Incidence and severity of adverse events (AEs) | Day 1 - Day 71.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of University of Science and Technology of China, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided